CLINICAL TRIAL: NCT03722511
Title: A Phase 2 Study Evaluating a Proprietary Amino Acid Based Medical Food (Enterade®) in Patients With Quality of Life Limiting Diarrhea Due to Carcinoid Syndrome and Other Neuroendocrine Tumors (NET).
Brief Title: Evaluating an Amino Acid Based Medical Food w/ Diarrhea in Carcinoid Syndrome & Other NETs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lowell Anthony, MD (Other)
Collaborators: Entrinsic Bioscience Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lowell Anthony, MD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-18-GI-101-EHS
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Neuroendocrine Tumors; Carcinoid Tumor of GI System; Diarrhea; Carcinoid Syndrome
Keywords: Enterade; Medical Food/Drink
MeSH Terms: conditions — Neuroendocrine Tumors; Diarrhea; Serotonin Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NET with carcinoid syndrome (Active Comparator): Participants with NET and carcinoid syndrome will be instructed to drink two 8 oz. bottles of Amino Acid Based Medical Food/Drink (Enterade®) per day.
  Interventions: Dietary Supplement: Amino Acid Based Medical Food/Drink
- NET w/o cardinoid syndrome (Active Comparator): Participants with NET w/o carcinoid syndrome will be instructed to drink two 8 oz. bottles of Amino Acid Based Medical Food/Drink (Enterade®) per day.
  Interventions: Dietary Supplement: Amino Acid Based Medical Food/Drink

INTERVENTIONS:
Dietary Supplement: Amino Acid Based Medical Food/Drink — Study Compound Enterade® is a medical food drink/beverage composed of a proprietary blend of electrolytes and amino acids.
  Other Names: Enterade®

SUMMARY:
Primary Objective:

To assess how an amino acid based medical food (Enterade®) helps maintain the intestine's ability to absorb and retain fluids, leading to a reduction in diarrhea due to Neuroendocrine Tumors (NET) and/or Carcinoid Syndrome. This improvement in the absorption will be assessed in part by evaluating changes in average daily stool frequency from baseline in patients receiving Enterade®. Each subject serves as his or her own control.

Secondary Objectives:

* To assess subject reported health-related quality of life in subjects before and after compound administration.
* To characterize the side effect profile and tolerability of Enterade® as measured by the number of total 8-oz Enterade® bottles consumed throughout the trial, and average drinks per day.
* To evaluate changes in serum electrolytes before and after administration of Eenterade®.
* To assess intravenous fluid requirement and/or hospitalization for dehydration secondary to diarrhea between control observation period and active Enterade® period.
* To evaluate difference in utilization of standard-of-care anti-diarrheal medications between control observation period and Enterade® period.
* To compare subjective feeling of bloating and flatulence before and after administration of Enterade®.
* To evaluate changes in patient weight before and after administration of Enterade®.

DETAILED DESCRIPTION:
This prospective, phase 2 study is to assess how Enterade® will affect patient-reported quality of life and intestinal absorption in patients with Carcinoid Syndrome and Neuroendocrine Tumors. The hypothesis is that Enterade® when combined with standard supportive care will improve patient-reported quality of life and help maintain the small bowel's ability to absorb and retain fluids, possibly leading to a reduction in diarrhea frequency.

* This is a non-randomized, supportive-care study.
* Potentially eligible patients will be screened in the University of Kentucky Markey Cancer Center clinics.
* During the screening visit, immediately after signing informed consent, the participant will be given both flavors of enterade® (original vanilla and refreshing orange) to test tolerability and taste.
* Eligible subjects will be given a stool diary and will be asked to document daily stool output (frequency and consistency of stool), use of anti-diarrheal medication and gastrointestinal discomforts (bloating, cramping).
* All lab and screening tests should be completed within 2 weeks prior to registration/initiation of study.
* The study is broken into 3 distinct segments and will apply to all enrolled participants: Baseline observation (Weeks 1-4), Enterade® administration period (4 weeks), Post-Enterade® Period (4 weeks).
* After relapse of diarrhea is documented or the 4 weeks of post-Enterade® observation are completed (whatever happens first), participants will be given the option to restart Enterade® for 1 additional month.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Participants must have histopathologically confirmed neuroendocrine tumor with 4 or more bowel movements per day on standard anti-diarrheal regimen (which may or may not include somatostatin analogs and telotristat), AND an elevated serum serotonin or plasma serotonin above the upper limit of normal per reference lab.
* Cohort 2: Participants who have histopathologically confirmed neuroendocrine tumor and have 4 or more bowel movements per day on standard anti-diarrheal regimen (which may or may not include somatostatin analogs and telotristat), but are below the cut-point for serotonin elevation.
* Age equal to or greater than 18 years old.
* ECOG performance status ≤2 (Karnofsky ≥60%)
* Ability to tolerate thin liquids by mouth at the time of enrollment.
* Ability to understand and the willingness to sign a written informed consent document.
* Subject who are willing to take enterade® as instructed will be eligible.

Exclusion Criteria:

* Known allergy to Stevia.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active Clostridium difficile infection or history of Clostridium difficile infection.
* Participants with active clostridium difficile infection will be ineligible for this study.
* Participants with a history of inflammatory bowel disease, irritable bowel syndrome, bariatric surgery and/or Celiac disease.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who have had enterade® within the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Effect of amino acids in tightening the intestinal barrier and protecting from antigenic translocation by evaluating plasma circulating cytokine levels in peripheral blood sample. | 56 days
  ELISA assays will be used to assess pro-inflammatory cytokines IL-1β, IL-6 and TNFα and serum endotoxin from blood samples collected.

SECONDARY OUTCOMES:
Evaluation of increased bacterial translocation and systemic inflammation. | 56 days
  Gut inflammation will be assessed through the analysis of fecal lactoferrin using stool specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Lowell Anthony, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No